CLINICAL TRIAL: NCT05433675
Title: A Single-center, Open-label, Single-dose, Randomized, 2-way Crossover Phase 1 Study in Healthy Adult Participants to Assess the Bioequivalence of the Dispersible Final Market Image (FMI) Macitentan Tablet (4 x 2.5 mg) and the Opsumit Tablet (10 mg) in Fasted Conditions
Brief Title: A Study of Two Macitentan Formulations in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR109185; 67896062PAH1010 (Other: Actelion); 2022-000262-17 (EudraCT Number)
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence AB (Experimental): Participants will receive single oral dose of macitentan formulated as dispersible final market image (FMI) in fasted conditions (test) (Treatment A) in Intervention Period 1 followed by a single oral dose of film-coated opsumit tablet in fasted conditions (reference) (Treatment B) in Intervention Period 2 on Day 1. There will be washout period of at least 10 days between two period.
  Interventions: Drug: Macitentan
- Treatment Sequence BA (Experimental): Participants will receive Treatment B in Intervention Period 1 followed Treatment A in Intervention Period 2 on Day 1. There will be washout period of at least 10 days between two period.
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan dispersible and film-coated tablets will be administered orally as per assigned treatment sequence.
  Other Names: Opsumit; ACT-064992; JNJ-67896062

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of macitentan on the primary pharmacokinetics (PK) parameters between the dispersible final market image (FMI) macitentan tablet and the opsumit tablet in healthy adult participants in fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical and surgical history performed at screening. If there are any abnormalities, they must be considered not clinically relevant and this determination must be recorded in the participant's source documents and initialed by the investigator
* Body weight not less than 50 kilograms (kg) and body mass index (BMI) within the range 18.5 - 30.0 kilogram per meter square (kg/m^2)(inclusive), at screening
* All women must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test at screening and must have a negative urine pregnancy test on Day -1 of each intervention period
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for a period of 30 days after the last study intervention intake
* Must sign an ICF indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study, before starting any screening activities

Exclusion Criteria:

* Known allergies, hypersensitivity, or intolerance to macitentan, fructose or drugs of the same class, or any excipients of the drug formulations
* History or clinical evidence of any disease or existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism, or excretion of the study intervention (appendectomy and herniotomy allowed, cholecystectomy not allowed)
* A history of repeated fainting due to cardiac cause, collapse, syncope, orthostatic hypotension, or vasovagal reactions
* Veins unsuitable for intravenous puncture on either arm (example, veins that are difficult to locate, access, or puncture, and veins with a tendency to rupture during or after puncture)
* Woman who is breastfeeding/pregnant at screening or plans to breastfeed/become pregnant throughout the study until 30 days after last study intervention intake

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of Macitentan | Predose up to 216 hours postdose (up to Day 10)
  Cmax is defined as maximum observed plasma analyte concentration of macitentan.
Area Under the Plasma Analyte Concentration Versus Time Curve From Time Zero To Time of the Last Quantifiable (Non-below Quantification Limit [Non-BQL]) Concentration (AUC [0-last]) of Macitentan | Predose up to 216 hours postdose (up to Day 10)
  AUC (0-last) is defined as area under the plasma analyte concentration versus time curve from time 0 to time of the last quantifiable (non-BQL) concentration of macitentan.
Area Under the Plasma Analyte Concentration-time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of Macitentan | Predose up to 216 hours postdose (up to Day 10)
  AUC (0-infinity) is defined as the area under the plasma analyte concentration-time curve from time 0 to infinite time of macitentan, calculated as the summation of AUC(0-last) and C(last)/lambda(z); where AUC(0-last) is area under the analyte concentration-time curve from time zero to last quantifiable time, Clast is the last observed measurable (non-BQL) plasma analyte concentration, and lambda(z) is apparent terminal elimination rate constant.

SECONDARY OUTCOMES:
Actual Sampling Time to Reach the Maximum Observed Plasma Analyte Concentration (Tmax) of Macitentan and Aprocitentan | Predose up to 216 hours postdose (up to Day 10)
  Tmax is defined as actual sampling time to reach the maximum observed plasma analyte concentration of macitentan and aprocitentan.
Last Observed Measurable (Non-BQL) Plasma Analyte Concentration (Clast) of Macitentan and Aprocitentan | Predose up to 216 hours postdose (up to Day 10)
  Clast is defined as last observed measurable (non-BQL) plasma analyte concentration of macitentan and aprocitentan.
Area Under the Plasma Analyte Concentration-time Curve from Time Zero to 72 Hours Postdose (AUC [0-72 Hours]) of Macitentan and Aprocitentan | Predose up to 0 to 72 hours postdose (up to Day 4)
  AUC (0-72 hours) is defined as area under the plasma analyte concentration-time curve from time 0 to 72 hours postdose of macitentan and aprocitentan calculated by linear-linear trapezoidal summation.
Apparent Terminal Elimination Half-life (t1/2) of Macitentan and Aprocitentan | Predose up to 216 hours postdose (up to Day 10)
  t1/2 is defined as apparent terminal elimination half-life of macitentan and aprocitentan, calculated as 0.693/lambda(z); where lambda(z) is apparent terminal elimination rate constant.
Apparent Terminal Elimination Rate Constant (Lambda[z]) of Macitentan and Aprocitentan | Predose up to 216 hours postdose (up to Day 10)
  Lambda(z) is defined as apparent terminal elimination rate constant of macitentan and aprocitentan, estimated by linear regression using the terminal log-linear phase of the log transformed concentration versus time curve.
Total Apparent Oral Clearance (CL/F) of Macitentan | Predose up to 216 hours postdose (up to Day 10)
  CL/F is defined as total apparent oral clearance of macitentan, calculated as dose/AUC (0-infinity).
Apparent Volume of Distribution (Vdz/F) of Macitentan | Predose up to 216 hours postdose (up to Day 10)
  Vdz/F of macitentan is defined as apparent volume of distribution of macitentan, calculated as dose/(Lambda[z]*AUC [0-infinity]).
Maximum Observed Plasma Analyte Concentration (Cmax) of Aprocitentan | Predose up to 216 hours postdose (up to Day 10)
  Cmax is defined as maximum observed plasma analyte concentration of aprocitentan.
Area Under the Plasma Analyte Concentration Versus Time Curve From Time Zero To Time of the Last Quantifiable (Non-BQL) Concentration (AUC [0-last]) of Aprocitentan | Predose up to 216 hours postdose (up to Day 10)
  AUC (0-last) is defined as area under the plasma analyte concentration versus time curve from time 0 to time of the last quantifiable (non-BQL) concentration of aprocitentan.
Area Under the Plasma Analyte Concentration-time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Aprocitentan | Predose up to 216 hours postdose (up to Day 10)
  AUC (0-infinity) is defined as the area under the plasma analyte concentration-time curve from time 0 to infinite time of aprocitentan, calculated as the summation of AUC(0-last) and C(last)/lambda(z); where AUC(0-last) is area under the analyte concentration-time curve from time zero to last quantifiable time, Clast is the last observed measurable (non-BQL) plasma analyte concentration, and lambda(z) is apparent terminal elimination rate constant.
Number of Participants with Serious Adverse Events (SAEs) | From screening to the last follow-up visit (up to 10 weeks)
  An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, or is an important medical event. An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product.
Number of Participants with Abnormalities in Physical Examination | Up to Day 10
  Number of participants with abnormalities in physical examination (including height and body weight) will be reported.
Number of Participants with Abnormalities in Vital Signs | Up to Day 10
  Number of participants with abnormalities in vital signs (including blood pressure, pulse/heart rate and oral temperature) will be reported.
Number of Participants with Abnormalities in Electrocardiogram (ECG) | Up to Day 10
  Number of participants with abnormalities in ECG will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to Day 10
  Number of participants with abnormalities in clinical laboratory tests (including hematology, serum chemistry, coagulation, serology and urinalysis) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (1):
- SGS Belgium NV, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency